CLINICAL TRIAL: NCT00308412
Title: Phase 1 Study to Determine the Safety, Infectivity, and Tolerability of Two Doses of Live Attenuated Recombinant Cold Passaged (cp) 45 Parainfluenza Type 3 Virus Vaccine, rHPIV3cp45, Lot PIV3 102A, Delivered as Nose Drops to Infants 6 to 12 Months of Age, and to HPIV3 Seronegative Infants and Children 6 to 36 Months of Age
Brief Title: Safety of and Immune Response to a Human Parainfluenza Virus Vaccine (rHPIV3cp45) in Healthy Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Ruth Karron, MD, Center for Immunization Research, Johns Hopkins School of Public Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CIR 215; CIR H.22.05.07.19.A1
Record Dates: First submitted 2006-03-28; First posted 2006-03-29 (Estimated); Last update posted 2010-07-16 (Estimated); Status verified 2010-07

CONDITIONS: Paramyxoviridae Infections; Virus Diseases
Keywords: Respiratory Tract Infection
MeSH Terms: conditions — Paramyxoviridae Infections; Virus Diseases; Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Two 10^5 PFU doses of rHPIV3cp45 vaccine given as nose drops to healthy infants and children aged 6 to 36 months of age. The two doses are given 4 to 10 weeks apart.
  Interventions: Biological: rHPIV3cp45
- 2 (Placebo Comparator): Two placebo vaccinations given as nose drops to healthy infants and children aged 6 to 36 months of age. The two doses are given 4 to 10 weeks apart.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: rHPIV3cp45 — Placebo for rHPIV3cp45 vaccine is 1X L-15.
  Arms: 1
Biological: Placebo — Placebo for rHPIV3cp45 vaccine
  Arms: 2

SUMMARY:
Human parainfluenza viruses (HPIVs) are a major health concern in infants and young children under 5 years of age, causing serious respiratory tract disease. The purpose of this study is to test the safety of and immune response to a new HPIV vaccine in healthy infants and children.

DETAILED DESCRIPTION:
HPIV type 3 (HPIV3) ranks second only to respiratory syncytial virus as the most important cause of bronchiolitis and pneumonia in infants less than 6 months of age. HPIV3 can cause severe disease in the first 2 years of life and is responsible for 11% of hospitalizations for respiratory diseases in children. This study will evaluate the safety and immunogenicity of a live recombinant attenuated intranasal HPIV3 vaccine, rHPIV3cp45.

This study will last for a maximum of 180 days. Infants will be enrolled into one of two study groups, Group 1 or Group 2. Depending on the study location, groups will enroll either sequentially or concurrently. Within each group, infants will be randomly assigned to receive 2 immunizations of rHPIV3cp45 or placebo. Immunizations will be given as nose drops. Immunizations will be given at study entry and approximately 4 to 10 weeks after study entry.

On the day of immunization, a physical exam, vital signs measurement, blood collection, and medical history will occur. Infants will be observed for 15 minutes after immunization for any immediate adverse effects. Parents or guardians will be given a thermometer to take with them and will be instructed on how to take their infant's temperature. They will be given the study schedule and will need to provide contact phone numbers so study personnel can contact them by phone during the days after immunization. Parents and guardians will be contacted by telephone on days without study visits, from Day 1 to Day 19 and on Day 180 after immunization, and asked about any illnesses or adverse effects they have observed in their immunized infants.

Parents or guardians will need to record their infant's temperature daily for at least the 17 days immediately following immunization. During this 17-day period, there will be at least 6 study visits associated with each immunization; visits will occur on the day of immunization and approximately 3, 7, 10, 14, and 17 days after immunization. At all study visits, infants will undergo a physical exam and vital signs measurement. Group 1 participants will also undergo a nasal wash for a viral culture. There will be additional follow-up visits occurring sometime between 28 and 70 days after the first dose and 28 to 35 days after the second dose; blood collection will occur at the follow-up visits. Additional visits may be required on selected days during the month after immunization. Infants who experience illness or side effects may be asked to return to the clinic for examination. Parents or guardians will be made aware of whether their infant received the HPIV vaccine or placebo 18 days after the second immunization or in the event of a lower respiratory tract illness.

ELIGIBILITY:
Inclusion Criteria for All Participants:

* Good general health
* Full term infant, born later than the 36th week of pregnancy
* Has received age-appropriate inactivated or subunit routine immunizations at least 2 weeks prior to study entry
* Has received age-appropriate live routine immunizations at least 4 weeks prior to study entry and at least 2 weeks for rotavirus vaccine
* Available for the duration of the trial
* Parent or guardian reachable by telephone for post-immunization contact
* Parent or guardian willing to provide informed consent
* For Group 2 participants, serum hemagglutination-inhibiting (HAI) titers to HPIV3 of or less than 1:8

Exclusion Criteria:

* Known or suspected impairment of immunologic functions. Infants who are HIV infected, who are bone marrow or solid organ transplant recipients, or who are using immunosuppressive therapy, including systemic corticosteroids, are excluded. Infants who are using topical steroids, topical antibiotic ointments and topical antifungal agents are not excluded.
* Major congenital malformations, including congenital cleft palate, cytogenetic abnormalities, or serious chronic disorders
* Previously received PIV3 vaccine
* Previous serious vaccine-associated adverse event or anaphylactic reaction
* Known hypersensitivity to any vaccine component
* Lung or heart disease, including reactive airway disease. Infants with clinically insignificant cardiac abnormalities are not excluded. Infants or children who wheezed once or received bronchodilator therapy once in the first year of life but who have not had any additional wheezing episodes or bronchodilator therapy for at least 12 months are not excluded.
* Born prematurely before the 37th week of pregnancy
* Member of a household containing immunocompromised individuals, pregnant caregivers, or infants less than 6 months of age
* Attends day care with infants less than 6 months of age
* Parent or guardian unable or unwilling to suspend daycare for 14 days following each immunization. More information on this criterion can be found in the protocol.
* Currently enrolled in another investigational drug or vaccine study

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2006-06; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Frequency of vaccine-related reactogenicity events (REs) that occur during the acute monitoring phase of the study | For 17 days after each dose
Proportion of infants that develop fourfold or greater rises in hemagglutination-inhibition (HAI) antibody titer following two doses of vaccine | Throughout study

SECONDARY OUTCOMES:
For the subset of infants enrolled in group 1 of the study (n=24), quantifying the amount of vaccine virus shed by each recipient | Throughout study
Assessment of the immunogenicity of a second dose of vaccine and the protection of the first dose against reinfection with the second dose | Throughout study
Determination of the number of vaccinated infants infected with rHPIV3cp45 | Throughout study
Determination of the number of vaccinated subjects infected with a second dose of rHPIV3cp45 vaccine | Throughout study
Determination of the phenotypic stability of vaccine virus shed | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Ruth A. Karron, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Center for Immunization Research, Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Background] Durbin AP, Karron RA. Progress in the development of respiratory syncytial virus and parainfluenza virus vaccines. Clin Infect Dis. 2003 Dec 15;37(12):1668-77. doi: 10.1086/379775. Epub 2003 Nov 20. PMID 14689350
- [Background] Greenberg HB, Piedra PA. Immunization against viral respiratory disease: a review. Pediatr Infect Dis J. 2004 Nov;23(11 Suppl):S254-61. doi: 10.1097/01.inf.0000144756.69887.f8. PMID 15577581
- [Background] Karron RA, Belshe RB, Wright PF, Thumar B, Burns B, Newman F, Cannon JC, Thompson J, Tsai T, Paschalis M, Wu SL, Mitcho Y, Hackell J, Murphy BR, Tatem JM. A live human parainfluenza type 3 virus vaccine is attenuated and immunogenic in young infants. Pediatr Infect Dis J. 2003 May;22(5):394-405. doi: 10.1097/01.inf.0000066244.31769.83. PMID 12792378
- [Background] Madhi SA, Cutland C, Zhu Y, Hackell JG, Newman F, Blackburn N, Murphy BR, Belshe RB, Karron RA, Deatly AM, Gruber WC, Bernstein DI, Wright PF. Transmissibility, infectivity and immunogenicity of a live human parainfluenza type 3 virus vaccine (HPIV3cp45) among susceptible infants and toddlers. Vaccine. 2006 Mar 20;24(13):2432-9. doi: 10.1016/j.vaccine.2005.12.002. Epub 2005 Dec 20. PMID 16406170
- [Background] Skiadopoulos MH, Surman SR, Riggs JM, Orvell C, Collins PL, Murphy BR. Evaluation of the replication and immunogenicity of recombinant human parainfluenza virus type 3 vectors expressing up to three foreign glycoproteins. Virology. 2002 May 25;297(1):136-52. doi: 10.1006/viro.2002.1415. PMID 12083844